CLINICAL TRIAL: NCT03831178
Title: Docosahexaenoic Acid (DHA) for Women With Breast Cancer in the Neoadjuvant Setting
Acronym: DHA-WIN
Status: Active, not recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: AHS Cancer Control Alberta (Other)
Collaborators: Canadian Institutes of Health Research (CIHR) (Other Government); University of Alberta (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: IIT-0005
Record Dates: First submitted 2019-01-14; First posted 2019-02-05 (Actual); Last update posted 2025-06-26 (Actual); Status verified 2025-06

CONDITIONS: Breast Cancer
MeSH Terms: conditions — Breast Neoplasms | interventions — Docosahexaenoic Acids

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- DHA (Experimental): Participants will take 11 capsules per day containing DHA-enriched triglyceride oil (1 g capsules containing at least 400 mg DHA) for a total of 5 g DHA/day divided into three times daily with meals or as tolerated.
  Interventions: Dietary Supplement: Docosahexaenoic acid (DHA)
- Placebo (Placebo Comparator): Participants will take 11 capsules per day containing corn/soy oil blend capsules divided into three times daily with meals or as tolerated.
  Interventions: Drug: Placebo oral capsule

INTERVENTIONS:
Dietary Supplement: Docosahexaenoic acid (DHA) — Participants will take 11 capsules of DHA oil for 12-18 weeks (84-126 days), beginning on day 1 of initial cycle of chemotherapy, and continuing for 4-6 cycles of chemotherapy prior to definitive breast surgery. Study will end when subject undergoes breast surgery.
  Arms: DHA
Drug: Placebo oral capsule — Participants will take 11 capsules of placebo (corn/soy oil blend) for 12-18 weeks (84-126 days), beginning on day 1 of initial cycle of chemotherapy, and continuing for 4-6 cycles of chemotherapy prior to definitive breast surgery. Study will end when subject undergoes breast surgery.
  Arms: Placebo

SUMMARY:
Docosahexaenoic acid (DHA) is an omega-3 long chain polyunsaturated fatty acid (n-3 LCPUFA). N-3 LCPUFA are essential fatty acids in the diet. The majority of n-3 LCPUFA in the diet is alpha-linolenic acid (ALA). While DHA can be synthesized from ALA and other n-3 LCPUFA in the body, endogenous synthesis is low. Consequently, the only way to significantly increase levels of DHA in tissues is by directly consuming this fatty acid. Common sources of DHA are fatty fish, fish oil and omega-3 supplements and fortified foods.

DHA is readily incorporated into membrane phospholipids and induces changes in the properties of the cell membrane including altered fluidity; permeability and membrane transport as well as activity of membrane bound receptors and enzymes.

It is well established that changes in membrane DHA has multiple effects in the body, including modulation of neurological, immune, and cardiovascular functions. In breast cancer, DHA increases sensitivity of breast cancer cells to different chemotherapeutic agents, and in animal models of breast cancer, dietary DHA decreases tumour growth. The investigator's preclinical studies demonstrate that DHA increases efficacy of both doxorubicin and docetaxel, two agents commonly used in the adjuvant setting for breast cancer treatment. Furthermore, DHA mitigates chemotherapy induced weight loss in mice, and reduces paclitaxel toxicities in breast cancer patients, strongly indicating that DHA protects against toxicity in normal tissues. Directly relevant to this study, increased DHA in breast adipose tissue correlates with improved response to chemotherapy, and increased dietary intake of n-3 LCPUFA, including DHA, results in increased DHA incorporation in breast adipose tissue. Lastly, in advanced metastatic breast cancer, DHA supplementation correlated with improved outcomes in a subset of patients. Consequently, the Investigators hypothesize that the therapeutic index (efficacy: toxicity ratio) will be improved with the addition of DHA. In this clinical trial, the Investigators will explore the benefit of DHA supplementation in combination with neoadjuvant chemotherapy in patients with early breast cancer.

RESEARCH QUESTION & OBJECTIVES: The Investigators propose to evaluate incorporation of DHA in women with breast cancer in treatment naïve patients in combination with chemotherapy, and assess potential benefit of DHA supplementation in breast cancer patients, using change in Ki67 labeling index (marker of proliferation) as a marker of efficacy. This study will further investigate the relationship between DHA in plasma phospholipids (as a potential biomarker of tumour incorporation) and effect on systemic immune function.

METHODS: Patients directed to receive chemotherapy will receive capsules, each containing a minimum of 400 mg of DHA in the form of DHA enriched triglyceride oil or placebo (corn/soy oil blend) to be taken orally (11 capsules/day, throughout day as preferred by participant) for a total of 5 g DHA or placebo, for 12-18 weeks (84-126 days) beginning at the start of the first cycle of chemotherapy, and continued throughout 4-6 cycles of chemotherapy (3 weeks/ cycle). DHA will be discontinued 21 days after the last administration of cytotoxic chemotherapy. Tumour biopsies at baseline and post surgical removal will be assessed for Ki67 status as well as for markers of apoptosis and stem cell presence (by immunohistochemistry). Blood samples taken at baseline prior to each round of chemotherapy will be assessed for immune markers and plasma phospholipid content.

ELIGIBILITY:
Inclusion Criteria:

1. Women with invasive (clinical stage I, II and III) breast cancer, for whom neoadjuvant systemic therapy with chemotherapy is recommended prior to surgery.
2. ECOG Performance status of 0 or 1.
3. Hematology and Biochemistry assessments (CBC and differential, PTT, PT/INR, AST, Alk Phos, Bilirubin, and Creatinine) within normal range unless determined not clinically significant by the qualified investigator.
4. Ability to take oral medications.
5. Adequate tissue specimen for diagnosis, biomarkers, and endpoint Ki67 assays.

Exclusion Criteria:

1. Patients undergoing surgery prior to chemotherapy.
2. Current or previous (within 2 months) daily use (>1 day/week) use of omega-3, fish oil, or other supplements or functional foods containing docosahexaenoic acid (at daily doses > 200 mg).
3. Known allergy to soy or corn.
4. Continued intake of supplements containing Vitamin C, Vitamin E or β-carotene exceeding the DRI, or other anti-oxidant supplements.
5. Symptomatic but untreated cholelithiasis.
6. History of deep venous thrombosis, active thrombophlebitis, pulmonary embolism, stroke, acute myocardial infarction, congestive cardiac failure, untreated hypertension, known inherited hypercoagulable disorder.
7. Diagnosis of any other malignancy within the previous year except for adequately treated basal cell or squamous cell skin cancer.
8. Medically documented history of a psychiatric disorder that would preclude consent
9. Partial or complete loss of vision or diplopia, from ophthalmic vascular disease.
10. Hypersensitivity to DHA or to any ingredient in the formulation or component of the container.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes
Enrollment: 76 (Actual)
Dates: Start 2019-08-28 (Actual); Primary Completion 2024-12-01 (Actual); Study Completion 2030-09 (Estimated)

PRIMARY OUTCOMES:
Percent change in Ki67 index from baseline to surgical excision. | Pre-intervention (on the baseline biopsy) and post- intervention (at the time of surgical excision).
  Ki67 will be measured by image analysis at baseline biopsy and at experimental end (surgical excision).

SECONDARY OUTCOMES:
Percent of DHA in plasma phospholipids between DHA and placebo arms. | At day 0 and day 20 of cycles 1 to 6 of chemotherapy (each cycle is 20 days).
  Changes in level of DHA incorporation in plasma phospholipids will be assessed to identify the range of DHA incorporation in this patient population. Fatty acid composition of plasma phospholipids will be measured after lipid extraction, phospholipid separation on thin layer chromatography followed by methylation and separation identification by gas-liquid chromatography.
Change in immune function (e.g. ability to produce IL-2 after stimulation) following DHA supplementation in combination with chemotherapy. | Baseline (within 21 days before cycle 1 of chemotherapy) and at the end of chemotherapy cycle 3 (each cyle is 20 days)
  Systemic immune function will be assessed on stored plasma by U-PLEX Biomarker Group 1 electrochemiluminescent multiplex assays (MesoScale Discovery).
Age of participants and other factors affecting DHA incorporation | Once participants undergo their breast surgery (within 3-6 weeks after the last chemotherapy cycle, each cycle is 20 days).
  If incorporation of DHA in plasma phospholipids is variable within the DHA treatment arm, possible factors that may influence incorporation (e.g. age of participants) will be explored between high and low incorporators.
Percent change on markers of apoptosis (e.g. caspase-3) following DHA or placebo supplementation. | Once participants undergo their breast surgery (within 3-6 weeks after the last chemotherapy cycle, each cycle is 20 days).
  Breast tissue from participants receiving DHA or placebo will be assessed for markers of apoptosis (e.g. caspase-3) by immunohistochemistry and calculated by image analysis.
Pathological complete response rate | Once participants undergo their breast surgery (within 3-6 weeks after the last chemotherapy cycle, each cycle is 20 days).
  Pathological complete response in resected breast tissue and all sampled axillary nodes will be assessed as absence of invasive cancer on haematoxylin and eosin evaluation as per standard of care.
Comparison of rate of chemotherapy associated grade 3 and 4 toxicities between treatment arms. | At day 20 of chemotherapy cycles 1 to 6 (each cycle is 20 days).
  Rate of chemotherapy associated grade 3 and 4 toxicities, and chemotherapy- associated hospitalizations will be compared between DHA and placebo arms.

CONTACTS AND LOCATIONS:
Overall Officials: John Mackey, MD, Principal Investigator — Cross Cancer Institute
Locations (1):
- Cross Cancer Institute, Edmonton, Alberta, Canada

IPD SHARING:
Plan to Share IPD: Yes
The Cross Cancer Institute and the University of Alberta encourages and supports the responsible and ethical sharing of data from clinical trials. The protocol and statistical analysis plan will be made available on Clinicaltrials.gov.
Supporting Information: Study Protocol, SAP, ICF
Time Frame: Documents will be published within 6 months after starting the trial.

REFERENCES:
- [Background] Newell M, Mackey JR, Bigras G, Alvarez-Camacho M, Goruk S, Ghosh S, Schmidt A, Miede D, Chisotti A, Postovit L, Baker K, Mazurak V, Courneya K, Berendt R, Dong WF, Wood G, Basi SK, Joy AA, King K, Meza-Junco J, Zhu X, Field C. Comparing docosahexaenoic acid (DHA) concomitant with neoadjuvant chemotherapy versus neoadjuvant chemotherapy alone in the treatment of breast cancer (DHA WIN): protocol of a double-blind, phase II, randomised controlled trial. BMJ Open. 2019 Sep 17;9(9):e030502. doi: 10.1136/bmjopen-2019-030502. PMID 31530611
- [Derived] Douglas CM, Newell M, Goruk S, Courneya KS, Ghosh S, Joy AA, Munhoz J, Field CJ. Exploratory outcomes of the DHA WIN randomized controlled trial: Supplementing women with docosahexaenoic acid did not reduce the impact of neoadjuvant breast cancer chemotherapy on quality of life or exercise behaviour. PLoS One. 2025 May 2;20(5):e0322178. doi: 10.1371/journal.pone.0322178. eCollection 2025. PMID 40315249